CLINICAL TRIAL: NCT06453759
Title: Thalamic Recordings in Children Undergoing SEEG
Acronym: TRICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23BI31
Record Dates: First submitted 2024-05-24; First posted 2024-06-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalamic SEEG (Experimental): The centromedian, anterior and pulvinar nuclei on each side will be chosen as target for new electrodes.
  Interventions: Procedure: Additional electrodes into bilateral anterior, centromedian and pulvinar thalamic nuclei

INTERVENTIONS:
Procedure: Additional electrodes into bilateral anterior, centromedian and pulvinar thalamic nuclei — The centromedian, anterior and pulvinar nuclei on each side will be chosen as target for new electrodes; up to 6 additional electrodes may be added but, where possible, existing electrode trajectories will be extended to facilitate recording.
  At the beginning of the recording process, usually within the first 24-48 hours of implantation, we will conduct 2 study-specific stimulation experiments:
  1. Single pulse electrical stimulation (SPES):
  2. N-of-1 trials of simulated DBS: We will simulate high (130Hz) and low (6Hz) frequency DBS currents from each pair of thalamic nuclei (always bilateral) and record spontaneous interictal neuronal activity in all other cortical contacts for 15 minutes. We will also record SPES from each of the cortical contacts.

SUMMARY:
Stereoelectroencephalography (SEEG) forms a key part of the pre-surgical evaluation in children who may be candidates for epilepsy surgery. It can help delineate the location of the putative epileptogenic zone, guiding further treatments including resective, disconnective and ablative epilepsy surgery techniques. However, less than 35% of children undergoing SEEG end up becoming seizure free following further treatment.

Open and closed loop stimulation of thalamic nuclei via deep brain stimulation (DBS) and responsive neurostimulation (RNS) are emerging treatment options for epilepsy. Thalamic target nuclei vary between studies and there are currently no gold standard personalised methods for choosing a target. This stems from the limited systematic neurophysiological recordings from thalamic nuclei; investigators currently do not understand the ictal and interictal thalamic signatures of involvement in epilepsy and do not understand how functional connectivity can be altered within and between patients.

In this prospective study, the investigators aim to recruit 30 patients undergoing SEEG as part of their pre-surgical evaluation for drug resistant epilepsy at Great Ormond Street Hospital over a period of 3 years. Once recruited, the investigators will target 3 nuclei bilaterally in each patient - the anterior, centromedian and pulvinar nuclei - using additional SEEG electrodes. Following clinical recording, the investigators will conduct two stimulation experiments, the first using single pulse electrical stimulation to measure effective connectivity between the thalamus and cortical regions and the second to study the effects of simulated DBS currents on cortical local field potential signatures.

This study will lay the foundation for a personalised approach to thalamic neuromodulation for drug-resistant epilepsy by identifying neurophysiological biomarkers of thalamic involvement in epilepsy, paving the way for closed loop neuromodulation strategies that aim to optimise response using these biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. All children undergoing SEEG as part of their pre-surgical evaluation at GOSH
2. Participants/parents/legal guardian provide informed consent for inclusion

Exclusion Criteria:

1) Lack of informed consent

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Ictal thalamic involvement | Hospital discharge (maximum one month from SEEG implantation)
  Experienced neurophysiologists will assess, during ictal activity, whether each of the nuclei are involved in the seizure and, if so, the latency between first cortical contact onset and thalamic nucleus onset.
Epileptogenicity index | Hospital discharge (maximum one month from SEEG implantation)
  We will quantify ictal involvement by measuring the epileptogenicity index in each nucleus.
Interictal power distribution | Hospital discharge (maximum one month from SEEG implantation)
  To assess interictal signatures, we will assess power at different frequencies in the nuclei using the 'fitting oscillations & one over f' (FOOOF) method.
Single pulse electrical stimulation (SPES): | Hospital discharge (maximum one month from SEEG implantation)
  We will systematically conduct SPES from all cortical and thalamic contacts and record responses in all other contacts. This measures the effective connectivity.

SECONDARY OUTCOMES:
Incidence of bleeding | Hospital discharge (maximum one month from SEEG implantation)
  Radiological evidence of bleeding or clinically new neurological symptoms during SEEG implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be allowed to be shared by our ethical approvals. We may make anonymised data available based on restrictions of ethical approvals.